CLINICAL TRIAL: NCT03021239
Title: Impact of Hemodynamic Ramp Test-Guided HVAD RPM and Medication Adjustments on Exercise Tolerance and Quality of Life: A Multicenter Study
Brief Title: Impact of Hemodynamic Ramp Test-Guided HVAD RPM and Medication Adjustments on Exercise Tolerance and Quality of Life
Acronym: Ramp-it-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1733
Record Dates: First submitted 2017-01-03; First posted 2017-01-13 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Continous Flow Left Ventricular Device
Keywords: Ramp Test; Continuous Flow -Left Ventricular Assist Device (CF-LVAD); LVAD Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) Echo Guided Testing - (Active Comparator): This testing uses echocardiography to create images of the heart and make measurements while gradually increasing the heart pump speed. The final pump speed and medical treatment are determined using the echo measurements. This will take about 45 minutes.
  Interventions: Procedure: Hemodynamic-Echo Ramp Testing -
- 2) Hemodynamic-Echo Ramp Testing - (Active Comparator): This testing is performed during a right heart catheterization procedure which provides hemodynamic measurements (pressure and blood flow) in addition to the echocardiography measurements. With this method, more echo images and measurements are taken. The final pump speed and medical treatment adjustments are made using the hemodynamic measurements as well as the information from the echo. This test will take about 1 hour and 45 minutes.
  Interventions: Procedure: Echo Guided Testing

INTERVENTIONS:
Procedure: Echo Guided Testing
  Arms: 2) Hemodynamic-Echo Ramp Testing -
Procedure: Hemodynamic-Echo Ramp Testing -
  Arms: 1) Echo Guided Testing -

SUMMARY:
The main purpose of this study is to compare Echo-guided testing to the Hemodynamic-Echo Ramp Tests to determine which method of testing provides better information for adjusting pump speed and medical treatment for Left Ventricular Assist Device (LVAD) patients. Better adjustments may provide better quality of life, exercise tolerance and reduced unwanted cardiac events over a 6-month period.

DETAILED DESCRIPTION:
All Left Ventricular Assist Device (LVAD)patients undergo testing to determine the best pumping speed for their Left Ventricular Assist Device (LVAD) and to gather measurements that help guide medical treatment. The testing uses echocardiography ("echo", ultrasound images of the heart) to create heart images and make measurements while gradually increasing the Left Ventricular Assist Device (LVAD) heart pump speed. Each time the pump speed is increased, images and measurements are taken. This is called a ramp test.

The ramp testing may also be performed during a right heart catheterization procedure. In a catheterization procedure, a doctor inserts a thin, flexible tube (catheter) into a vein or artery in the upper leg (groin), arm or neck and guides it to the heart using X-ray imaging. Doctors normally perform this procedure to measure the pressure and blood flow in the heart (otherwise called hemodynamic measurements). If the ramp testing is performed during this procedure, then the doctors have additional measurements to consider before choosing a final speed for the Left Ventricular Assist Device (LVAD) pump and appropriate medical treatment.

All of the procedures in this study are considered standard of care. The research part is randomly assigning the subject to one of the two methods of testing in this study. Subjects have a 50/50 chance of being in either testing group.

Baseline Visit (1 - 3 months after Left Ventricular Assist Device (LVAD) implant)

The following will be performed:

* Subjects will be asked to sign this consent form.
* Physical exam with an assessment of heart failure symptoms, and medical history will be recorded
* Routine blood tests (about 1 tablespoon will be drawn)
* Subjects will be randomly assigned to one of the two testing groups. If there is time, the ramp test can be performed at this visit, but usually it will be scheduled to occur a different day in about 1 to 4 weeks.
* 6 Minute Walk Test. This test measures how far the subject can walk in 6 minutes. If needed, this can be completed the day of the ramp test.
* Subjects will be asked to complete a questionnaire about their current quality of life. This will take about 10 minutes. If needed, this can be completed the day of the ramp test.

Ramp Testing Groups:

1. Echo Guided Testing - This testing uses echocardiography to create images of the heart and make measurements while gradually increasing the heart pump speed. The final pump speed and medical treatment are determined using the echo measurements. This will take about 45 minutes.

   OR
2. Hemodynamic-Echo Ramp Testing - This testing is performed during a right heart catheterization procedure which provides hemodynamic measurements (pressure and blood flow) in addition to the echocardiography measurements. With this method, more echo images and measurements are taken. The final pump speed and medical treatment adjustments are made using the hemodynamic measurements as well as the information from the echo. This test will take about 1 hour and 45 minutes.

6 Months after Baseline Visit

The following will be performed:

* Physical exam with an assessment of heart failure symptoms, and medical history will be recorded
* Routine blood tests (about 1 tablespoon will be drawn)
* 6 Minute Walk Test. This test measures how far the subject can walk in 6 minutes.
* Subjects will be asked to complete a questionnaire about their current quality of life. This will take about 10 minutes.
* All subjects will undergo a Hemodynamic-Echo Ramp Test at 6 months after the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. Newly implanted HVAD
3. HVAD support anticipated for at least 6 months
4. Patient is ambulatory and discharged from hospital without inotropes
5. Patient is between 1 and 3 months post implant
6. Patient has not had a right heart catheterization since discharged from HVAD implantation hospitalization

Exclusion Criteria:

1. The current HVAD is a replacement device
2. Patients currently has Right Ventricle (RV) failure requiring home inotropes
3. Inability to preformed right heart cath
4. Inadequate echocardiographic windows

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Clinical parameters most likely to be impacted by hemodynamic-echo ramp tests | 6 Months
  6 Walk Test
Heart Failure Readmission | 6 Months
  Composite end-point of heart failure readmission.
Quality of Life: Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 Months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) a summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains in which scores are transformed to a range of 0-100.
New York Heart Association (NYHA) Class | 6 Months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UC San Diego Medical Center, San Diego, California
  - Stanford Medical Center, Stanford, California
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uriel N, Burkhoff D, Rich JD, Drakos SG, Teuteberg JJ, Imamura T, Rodgers D, Raikhelkar J, Vorovich EE, Selzman CH, Kim G, Sayer G. Impact of Hemodynamic Ramp Test-Guided HVAD Speed and Medication Adjustments on Clinical Outcomes. Circ Heart Fail. 2019 Apr;12(4):e006067. doi: 10.1161/CIRCHEARTFAILURE.119.006067. PMID 30946600